CLINICAL TRIAL: NCT04520685
Title: CAnnabidiol Study in Children With Autism Spectrum DisordEr (CASCADE): A Double-Blind, Placebo-Controlled Study to Investigate Efficacy and Safety of Cannabidiol in Children and Adolescents With Autism
Brief Title: CASCADE: CAnnabidiol Study in Children With Autism Spectrum DisordEr
Acronym: CASCADE
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 19-2168
Record Dates: First submitted 2020-07-29; First posted 2020-08-20 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-05

CONDITIONS: Autism Spectrum Disorder
Keywords: CBD; cannabidiol; ASD; autism spectrum disorder; autism
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — Cannabidiol

STUDY DESIGN:
Intervention Model Description: For this study, participants will be randomly assigned to one of the following groups:
  1. Group A will receive cannabidiol for the first 12 weeks of the study and placebo for the last 15 weeks.
  2. Group B will receive placebo for the first 15 weeks of the study and cannabidiol for the last 12 weeks
  3. Group C will receive cannabidiol throughout the entire 27 weeks of treatment
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Arm 1: 12 weeks of study drug then 15 weeks of placebo (Experimental): Subjects in this group will receive cannabidiol for the first 12 weeks of the study and placebo for the last 15 weeks.
  Interventions: Drug: Oral cannabidiol 100mg/mL; Drug: Placebo
- Arm 3: 15 weeks of placebo then 12 weeks of study drug (Experimental): Subjects in this group will receive placebo for the first 15 weeks of the study and cannabidiol for the last 12 weeks.
  Interventions: Drug: Oral cannabidiol 100mg/mL; Drug: Placebo
- Arm 3: 27 weeks of study drug (Experimental): Subjects in this group will receive cannabidiol throughout the entire 27 weeks of treatment.
  Interventions: Drug: Oral cannabidiol 100mg/mL

INTERVENTIONS:
Drug: Oral cannabidiol 100mg/mL — In Arm 1, patients will begin CBD in period 1 and receive placebo in period 2. In Arm 2, patients will begin placebo in period 1 and receive CBD in period 2. In Arm 3, patients will receive CBD for the entire 27 week study duration without washout. Each study period is 12 weeks and dose will be titrated up for 1 week at the beginning of a treatment period and titrated down for 1 week at the end of a treatment period, with a two week placebo washout between periods for Arms 1 and 2. The titration dose will be 5mg/kg/day and the treatment dose will be 10mg/kg/day.
Drug: Placebo — In Arm 1, patients will begin CBD in period 1 and receive placebo in period 2. In Arm 2, patients will begin placebo in period 1 and receive CBD in period 2. In Arm 3, patients will receive CBD for the entire 27 week study duration without washout. Each study period is 12 weeks and dose will be titrated up for 1 week at the beginning of a treatment period and titrated down for 1 week at the end of a treatment period, with a two week placebo washout between periods for Arms 1 and 2. The titration dose will be 5mg/kg/day and the treatment dose will be 10mg/kg/day.
  Arms: Arm 1: 12 weeks of study drug then 15 weeks of placebo; Arm 3: 15 weeks of placebo then 12 weeks of study drug

SUMMARY:
This is a randomized, placebo-controlled study but all study participants will receive the active study medication at some point during the study for at least 12 weeks, and some children with receive CBD for the entire study.

DETAILED DESCRIPTION:
Autism spectrum disorder (ASD) is a relatively common neurodevelopmental disorder manifest by social communication deficits and restricted and repetitive interests. Individuals with ASD often have behavioral issues and psychiatric comorbidities which can be very hard to manage. Currently, there are only two FDA approved medications (aripiprazole and risperidone) for the treatment of irritability in ASD. Both medications have the potential for side effects and are not tolerated in all children with ASD. Anecdotal and some preliminary studies suggest that cannabidiol (CBD), a non-psychoactive cannabinoid in the marijuana plant, may lead to improvements in symptoms of ASD including irritability, aggressive behaviors, and anxiety.

In this study the investigators will test whether CBD leads to differences in behaviors commonly associated with ASD. The main behavioral problems investigators will study are irritability and aggressive behavior. This study will also measure changes in other behaviors seen in ASD such as anxiety, social interaction difficulties, repetitive behaviors, attentional problems, hyperactivity, repetitive behaviors, and quality of life. Study investigators will also test whether there are any important side effects of CBD in children and adolescents with ASD.

ELIGIBILITY:
Inclusion Criteria:

* Male or female children and adolescents aged 5-17 years, inclusive, at the time of screening.
* Judged by the investigator to be in good health at screening based upon the results of a medical history, physical examination, 12-lead ECG, and clinical laboratory test results.
* Patients must have a previous documented diagnosis of ASD by a medical or psychological professional.
* Patients must be assessed by the Investigator as being moderately to severely impacted due to ASD
* Patients who are taking psychotropic medication(s) should be on a stable regimen of no more than 2 medications for at least 4 weeks preceding study Screening and must maintain that regimen throughout the study. Psychotropic medications include (but are not limited to) antipsychotics, antidepressants, mood stabilizers, anxiolytics, and ADHD medications.
* Patients with a history of seizure disorders must currently be receiving treatment with a stable regimen of one or two AEDs, or must be seizure-free for 1 year if not currently receiving AEDs.
* Patients with seizures should be on a stable regimen for the 3 months preceding study enrollment of no more than 2 of the permitted anti-epileptic drugs (AEDs). Patients must remain on a stable AED dose throughout the study.
* If patients are receiving non-pharmacological educational, behavioral, and/or dietary interventions or therapies, they must be stable and have been doing so for 2 months prior to screening. Changes with school breaks are expected and do not apply.
* Patients must have a BMI of between 12-32 kg/m2 (inclusive).
* Females of childbearing potential and must have a negative serum pregnancy test at the Screening Visit and a negative urine pregnancy test at all designated visits.
* Patients/caregivers agree to abide by all study restrictions and comply with all study procedures.
* Parents/caregivers must be able to read and respond to questions and questionnaires in English.
* Patients/caregivers must be adequately informed of the nature and risks of the study and give written informed consent prior to screening.
* Parents/caregiver(s) must provide written consent to assist in study drug administration.
* In the Investigator's opinion, patients/caregivers are reliable and willing and able to comply with all protocol requirements and procedures (including scheduled visits and confinement periods).

Exclusion Criteria:

* Adolescent females who are pregnant, nursing, or planning a pregnancy. Females of childbearing potential and male patients with a partner of childbearing potential who are unwilling or unable to use standard acceptable methods of contraception (including abstinence, hormonal contraception, diaphragm, cervical cap, vaginal sponge, condom, or intrauterine device) for the duration of the study and for 1 month after the last dose of study medication.
* History of significant allergic condition, significant drug-related hypersensitivity, or allergic reaction to any compound or chemical class related to CBD (Epidiolex) or its ingredients.
* Exposure to any investigational drug or device < 30 days prior to screening, or plans to take another investigational drug at any time during the study.
* Use of any THC or CBD-containing product within 4 weeks of Screening Visit, planned use during the study, or positive THC urine test at screening.
* Patient is using the following medications: clobazam (Onfi, Frisium), felbamate (Felbatol), vigabatrin (Sabril), or everolimus (Afinitor).
* Plan to initiate or change pharmacologic or non-pharmacologic interventions during the course of the study.
* Patient has ALT, AST, total bilirubin, or creatinine levels ≥ 2 times the ULN, alkaline phosphatase levels ≥ 3 times the ULN, or Hct <1.2 times the LLN as determined from screening safety laboratories.
* Severe or unstable symptoms of ASD that may interfere with the study outcome evaluations and interpretation of results.
* Suffering from acute or progressive neurological disease, psychosis, schizophrenia or any psychiatric disorder or severe psychiatric abnormalities that are likely to require changes in drug therapy or interfere with the objectives of the study or the ability to adhere to protocol requirements.
* Has suspected or confirmed cardiovascular disease.
* History of treatment for, or evidence of, drug or alcohol abuse within the past year.

Ages: 5 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 86 (Actual)
Dates: Start 2021-12-15 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist- 2nd Edition (ABC-2): Irritability subscale raw score | Baseline to Week 12
  The Aberrant Behavior Checklist- 2nd Edition (ABC-2) is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The ABC-2 is a 58-item questionnaire and measures domains of Irritability, Lethargy/Social Withdrawal, Stereotypic Behavior, Hyperactivity/noncompliance, and Inappropriate Speech. Behaviors are assessed using a 4-point Likert scale. Scores range from "not at all a problem" (0) to "the problem is severe in degree" (3). The Irritability subscale range is from 0 to 45.

SECONDARY OUTCOMES:
Aberrant Behavior Checklist- 2nd Edition (ABC-2): Lethargy/Social Withdrawal subscale | Baseline to Week 12
  The Aberrant Behavior Checklist- 2nd Edition (ABC-2) is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The ABC-2 is a 58-item questionnaire and measures domains of Irritability, Lethargy/Social Withdrawal, Stereotypic Behavior, Hyperactivity/noncompliance, and Inappropriate Speech. Behaviors are assessed using a 4-point Likert scale. Scores range from "not at all a problem" (0) to "the problem is severe in degree" (3). The Lethargy/Social Withdrawal subscale range is from 0 to 48.
Aberrant Behavior Checklist- 2nd Edition (ABC-2): Stereotypic Behavior subscale | Baseline to Week 12
  The Aberrant Behavior Checklist- 2nd Edition (ABC-2) is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The ABC-2 is a 58-item questionnaire and measures domains of Irritability, Lethargy/Social Withdrawal, Stereotypic Behavior, Hyperactivity/noncompliance, and Inappropriate Speech. Behaviors are assessed using a 4-point Likert scale. Scores range from "not at all a problem" (0) to "the problem is severe in degree" (3). The Stereotypic Behavior subscale range is from 0 to 21.
Aberrant Behavior Checklist- 2nd Edition (ABC-2): Inappropriate Speech subscale | Baseline to Week 12
  The Aberrant Behavior Checklist- 2nd Edition (ABC-2) is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The ABC-2 is a 58-item questionnaire and measures domains of Irritability, Lethargy/Social Withdrawal, Stereotypic Behavior, Hyperactivity/noncompliance, and Inappropriate Speech. Behaviors are assessed using a 4-point Likert scale. Scores range from "not at all a problem" (0) to "the problem is severe in degree" (3). The Inappropriate Speech subscale range is from 0 to 12.
Aberrant Behavior Checklist- 2nd Edition (ABC-2): Hyperactivity/Noncompliance subscale | Baseline to Week 12
  The Aberrant Behavior Checklist- 2nd Edition (ABC-2) is a standard parent/caregiver reported behavioral outcome measure for use in developmental disability clinical trials. The ABC-2 is a 58-item questionnaire and measures domains of Irritability, Lethargy/Social Withdrawal, Stereotypic Behavior, Hyperactivity/noncompliance, and Inappropriate Speech. Behaviors are assessed using a 4-point Likert scale. Scores range from "not at all a problem" (0) to "the problem is severe in degree" (3). The Hyperactivity/Noncompliance subscale range is from 0 to 48.
Anxiety, Depression, and Mood Scale (ADAMS): Total Score | Baseline to Week 12
  The Anxiety, Depression, and Mood Scale (ADAMS) is a 28-item parent-report scale designed for individuals with disabilities to measure domains of anxiety (range 0 - 21), depression (range 0 - 21), hyperactivity (range 0 - 15), social avoidance (range 0 - 21), and obsessive/compulsive behavior (range 0 - 9). The total score is the sum of all items (range 0 - 87). Items are rated on a scale of "not a problem" (0) to "severe problem" (3).
Anxiety, Depression, and Mood Scale (ADAMS): General Anxiety subscale | Baseline to Week 12
  The Anxiety, Depression, and Mood Scale (ADAMS) is a 28-item parent-report scale designed for individuals with disabilities to measure domains of anxiety (range 0 - 21), depression (range 0 - 21), hyperactivity (range 0 - 15), social avoidance (range 0 - 21), and obsessive/compulsive behavior (range 0 - 9). The total score is the sum of all items (range 0 - 87). Items are rated on a scale of "not a problem" (0) to "severe problem" (3).
Anxiety, Depression, and Mood Scale (ADAMS): Social Avoidance subscale | Baseline to Week 12
  The Anxiety, Depression, and Mood Scale (ADAMS) is a 28-item parent-report scale designed for individuals with disabilities to measure domains of anxiety (range 0 - 21), depression (range 0 - 21), hyperactivity (range 0 - 15), social avoidance (range 0 - 21), and obsessive/compulsive behavior (range 0 - 9). The total score is the sum of all items (range 0 - 87). Items are rated on a scale of "not a problem" (0) to "severe problem" (3).
Social Responsiveness Scale - 2nd Edition (SRS-2): total T-score | Baseline to Week 12
  The Social Responsiveness Scale - 2nd Edition (SRS-2) is a standardized questionnaire that provides T-scores in domains of social communication, social motivation, social cognition, and restrictive/repetitive behaviors. The SRS-2 Total T-score ranges from 30 to ≥90 with higher scores indicating greater deficiencies in reciprocal social behavior.
Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) scale | Baseline to Week 12
  The Ohio Autism Clinical Impressions Scale - Severity (OACIS-S) is a 10-item, clinician completed measures based upon interview and/or observation. The OACIS-S assesses severity in domains of social interaction, aberrant behavior (including irritability and aggressive behavior), repetitive or ritualistic behavior, verbal communication, nonverbal communication skills, hyperactivity and inattention, anxiety and fearfulness, sensory sensitivities, restricted and narrow interests, and a global rating of autism severity. A 7-point Likert scale is used with scores ranging from "normal" (1) to "among the most severe" (7).
Ohio Autism Clinical Impressions Scale - Improvement (OACIS-I) scale | Baseline to Week 12
  The Ohio Autism Clinical Impressions Scale - Improvement (OACIS-I) is a 10-item, clinician completed measures based upon interview and/or observation. The OACIS-I assesses improvement in domains of social interaction, aberrant behavior (including irritability and aggressive behavior), repetitive or ritualistic behavior, verbal communication, nonverbal communication skills, hyperactivity and inattention, anxiety and fearfulness, sensory sensitivities, restricted and narrow interests, and a global rating of autism severity. A 7-point Likert scale is used with scores ranging from "very much improved" (1) to "very much worse" (7).
Autism Screening Instrument for Educational Planning - 3rd Edition (ASIEP - 3): Interaction Assessment Autism Interaction Score | Baseline to Week 12
  The Autism Screening Instrument for Educational Planning - 3rd Edition (ASIEP-3) is a 12-minute play-based assessment that evaluates social interactions and social responses. Videos of the session are coded for interactions, social avoidance, and negative behaviors (self-stimulatory, aggression). The vocal behavior is also coded as a separate domain to provide a sample of language function.
Repetitive Behavior Scale - Revised (RBS-R) | Baseline to Week 12
  The Repetitive Behavior Scale - Revised (RBS-R) is a caregiver-completed, 43-item questionnaire assessing repetitive behaviors with 6 subscales: stereotyped (range 0 - 27), ritualistic/sameness (range 0 - 36) , self-injurious (range 0 - 24), compulsive (range 0 - 18), and restricted (range 0 - 9). The total score ranges from 0 to 129, with a higher score indicating more significant problems with repetitive behaviors. Repetitive Behaviors are assessed using a 4-point Likert scale. Scores range from "behavior does not occur" (0) to "behavior occurs and is a severe problem" (3).
Brief Rating Inventory of Executive Functioning - 2nd edition (BRIEF-2): Global Executive Functioning Score | Baseline to Week 12
  The Brief Rating Inventory of Executive Functioning - 2nd edition (BRIEF-2) is a standardized rating scale that measures domains of executive functioning, including behavior regulation (inhibition, self-monitoring), emotional regulation (shifting, emotional control), and cognitive regulation (initiation, working memory, plan/organize, task monitoring, and organization of materials). It is made up of 63 items with three answer options (1 = Never; 2= Sometimes; 3=Often). Each item on the parent form is scored 1-3 (1 = Never; 2 = Sometimes; 3 = Often), yielding a raw score of the global scale range from 63 to 189. T scores (M = 50, SD = 10) are used to interpret the level of executive functioning. T-score range is 0-100, and higher scores are indicative of more severe deficiency - 65 or higher is considered to be in the "clinically significant" range.
Brief Rating Inventory of Executive Functioning - 2nd edition (BRIEF-2): ADHD score | Baseline to Week 12
  The Brief Rating Inventory of Executive Functioning - 2nd edition (BRIEF-2) is a standardized rating scale that measures domains of executive functioning, including behavior regulation (inhibition, self-monitoring), emotional regulation (shifting, emotional control), and cognitive regulation (initiation, working memory, plan/organize, task monitoring, and organization of materials). It is made up of 63 items with three answer options (1 = Never; 2= Sometimes; 3=Often). For the ADHD score, 18 items on the BRIEF-2 that correlate with clinical criteria for a diagnosis of ADHD each receive a score from 1-3 (1 = Never; 2 = Sometimes; 3 = Often). These items are summed and produce a range from 18-54, with higher values indicating more ADHD symptoms.
Brief Rating Inventory of Executive Functioning - 2nd edition (BRIEF-2): Index scores | Baseline to Week 12
  The Brief Rating Inventory of Executive Functioning - 2nd edition (BRIEF-2) is a standardized rating scale that measures domains of executive functioning, including 3 index scores of behavior regulation (inhibition, self-monitoring), emotional regulation (shifting, emotional control), and cognitive regulation (initiation, working memory, plan/organize, task monitoring, and organization of materials). It is made up of 63 items with three answer options (1 = Never; 2= Sometimes; 3=Often). Each item on the parent form is scored 1-3 (1 = Never; 2 = Sometimes; 3 = Often), yielding a raw score of the global scale range from 63 to 189. T scores (M = 50, SD = 10) are used to interpret the level of executive functioning. T-score range is 0-100, and higher scores are indicative of more severe deficiency - 65 or higher is considered to be in the "clinically significant" range.
Sleep Clinical Global Impressions - Severity Scale (Sleep CGI-S) | Baseline to Week 12
  The Sleep Clinical Global Impressions - Severity Scale (Sleep CGI-S) is a clinician completed measure based upon interview which assesses severity in domains of ability to fall asleep and remain sleeping independently, bedtime resistance; sleep onset delay; night awakening; caregiver satisfaction with their child's current sleep patterns; family functioning, as affected by their child's current sleep patterns. A 7-point Likert scale is used for each domain with scores ranging from "no concerns"/"does not occur" (1) to "Among the worst" (7).
Sleep Clinical Global Impressions - Improvement Scale (Sleep CGI-I) | Baseline to Week 12
  The Sleep Clinical Global Impressions - Improvement Scale (Sleep CGI-I) is a clinician completed measure based upon interview which assesses improvement in domains of ability to fall asleep and remain sleeping independently, bedtime resistance; sleep onset delay; night awakening; caregiver satisfaction with their child's current sleep patterns; family functioning, as affected by their child's current sleep patterns. A 7-point Likert scale is used for each domain with scores ranging from "very much improved" (1) to "very much worse" (7).
Autism Family Experience Questionnaire (AFEQ) | Baseline to Week 12
  The Autism Family Experience Questionnaire (AFEQ) is a 48-item questionnaire that measures family quality of life with domains of experience of being a parent (range 13 - 65), family live (range 9 - 45), child development and social relationships (range 14 - 70), and child's feelings and behavior (range 12 - 60). The sum of all domains gives the total score (range 48 - 240). Each question is assessed using a 5-point Likert scale. Scores range from "always" (1) to "never" (5)". For the total score and the domain scores a higher score indicates a lower outcome.
NIH Toolbox Scales: Satisfaction with Social Roles and Activities - Short Form 4a | Baseline to Week 12
  National Institutes of Health Patient Reported Outcome Measures Information System (NIH PROMIS) will be used to quantify psychological wellbeing and quality of life through self-report and/or parent proxy report. Satisfaction with Social Roles and Activities - Short Form 4a assesses satisfaction with performing one's usual social roles and activities and uses a 5-point Likert scale with scores ranging from "not at all" (1) to "very much" (5). The sum of all scores yields a total raw score (range 4 - 20) with higher scores indicating a greater level of satisfaction. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10.
NIH Toolbox Scales: Life Satisfaction - Short Form 8b | Baseline to Week 12
  National Institutes of Health Patient Reported Outcome Measures Information System (NIH PROMIS) will be used to quantify psychological wellbeing and quality of life through self-report and/or parent proxy report. Life Satisfaction - Short Form 8b assesses an individual's cognitive evaluation of life experiences and whether one likes his/her life or not. Each question is scored using a 5-point Likert scale with scores ranging from "not at all" (1) to "very much" (5). The sum of all scores yields a total raw score (range 8 - 40) with higher scores indicating a greater level of satisfaction. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10.
NIH Toolbox Scales: Positive Affect - Short Form 4a | Baseline to Week 12
  National Institutes of Health Patient Reported Outcome Measures Information System (NIH PROMIS) will be used to quantify psychological wellbeing and quality of life through self-report and/or parent proxy report. Positive Affect - Short Form 41 assesses momentary positive or rewarding affective experiences, such as feelings and mood associated with pleasure, joy, happiness, and excitement. Each question is scored using a 5-point Likert scale with scores ranging from "not at all" (1) to "very much" (5). The sum of all scores yields a total raw score (range 4 - 20) with higher scores indicating a greater level of positive affect. The final score is represented by the T-score, a standardized score with a mean of 50 and a standard deviation (SD) of 10.
Pediatric Quality of Life Inventory (PedsQL) - Core Scale | Baseline to Week 12
  The Pediatric Quality of Life Inventory (PedsQL) - Core Scale is a 23-item caregiver questionnaire to evaluate overall quality of life (QOL) in domains of physical functioning, emotional functioning, social functioning, and school functioning. A 5-point Likert scale is used with responses ranging from "Never" (0) to "Almost Always" (4). Items are reversed scored and transformed to a 0 - 100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. The total score is the sum of all the items over the number of items answered with higher scores indicating better health-related quality of life (HRQoL).
Pediatric Quality of Life Inventory (PedsQL) - Cognitive Functioning Scale | Baseline to Week 12
  The Pediatric Quality of Life Inventory (PedsQL) - Cognitive Scale is a 6-item caregiver questionnaire to evaluate an individual's mental abilities including learning, thinking, remembering and attention . A 5-point Likert scale is used with responses ranging from "Never" (0) to "Almost Always" (4). Items are reversed scored and transformed to a 0 - 100 scale as follows: 0=100, 1=75, 2=50, 3=25, and 4=0. The total score is the sum of all the items over the number of items answered with higher scores indicating lower problems.

OTHER OUTCOMES:
AutismEyes Eyetracking system Autism Symptoms Index (ASI) | Baseline to Week 12
  AutismEYES is an eye tracking device that is an objective, quantitative set of measurements that has been validated as both a diagnostic tool and measure of severity in children with ASD.
Telehealth Functional Behavior Analysis (Tele-FBA) | Baseline to Week 12
  A Functional Analysis (FA) evaluates variables that influence the occurrence of problem behavior by directly evaluating behaviors in natural settings.
Autism Screening Instrument for Educational Planning- 3rd Edition Sample of Vocal Behavior (ASIEP-3 SVB) Vocalization Score | Baseline to Week 12
  The Autism Screening Instrument for Educational Planning - 3rd Edition (ASIEP-3) is a 12-minute play-based assessment that evaluates social interactions and social responses. Videos of the session are coded for interactions, social avoidance, and negative behaviors (self-stimulatory, aggression). The vocal behavior is also coded as a separate domain to provide a sample of language function.
Parent/Caregiver Improvement Scale | Baseline to Week 12
  The Parent/Caregiver Improvement Scale is caregiver-completed questionnaire that assesses improvement in domains of communication skills, social skills, daily living skills and overall behavioral symptoms. A 7-point Likert scale is used for each domain with scores ranging from "very much improved" (1) to "very much worse" (7).

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Hospital Colorado, Aurora, Colorado, United States

REFERENCES:
- [Derived] Sannar EM, Winter J, Franke RK, Werner E, Rochowiak R, Romani PW, Miller OS, Semmler N, Bainbridge JL, Natvig C, Mikulich-Gilbertson SK, Tartaglia NR. Cannabidiol for treatment of irritability and aggressive behavior in children and adolescents with autism spectrum disorder: background and methods of the cannabidiol study in children with autism spectrum disorder study. Int J Clin Trials. 2025 Jan-Mar;12(1):29-37. doi: 10.18203/2349-3259.ijct20250131. Epub 2025 Jan 28. PMID 41103807
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711